CLINICAL TRIAL: NCT04248023
Title: Practice Facilitation to Promote Evidence-based Screening and Management of Unhealthy Alcohol Use in Primary Care
Brief Title: Screening and Management of Unhealthy Alcohol Use in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HM20016728; 1R18HS027077-01 (AHRQ)
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Alcohol Drinking; Alcohol Abuse; Alcohol Use Disorder
Keywords: Alcohol Misuse; Alcohol Abuse; Practice Facilitation; Motivational Interviewing; Preventive Services
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Intervention Model Description: This study is a practice level randomized controlled trial. 125 practices across Virginia will receive the intervention (practice facilitation to enhance screening and treatment of unhealthy alcohol use (UAU)) or act as a control group (will receive practice facilitation at 3 month lag behind intervention groups.) The investigators will survey 60 patients from each practice at three time intervals to evaluate the current state and what changes are implemented and reported over the course of the study. An additional 60 patient chart review from each practice will be preformed. The investigators will use an implementation-effectiveness design to measure outcomes. Effectiveness outcomes include increased screening rate of patients; increased treatment of any kind for patients with UAU; and reduction of UAU. Implementation outcomes will include the barriers and facilitators to screening and evaluating for UAU.
Masking Description: Based on the intervention of practice facilitation, it is not able to blind practices or clinicians from the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Practices (Experimental): Intervention practices will work with a practice facilitator to make practice specific changes to address unhealthy alcohol use.
  Interventions: Behavioral: Practice Facilitation
- Control Practices (No Intervention): Control practices will continue to screening and address unhealthy alcohol use based on their existing practice patterns.

INTERVENTIONS:
Behavioral: Practice Facilitation — A practice facilitator will be assigned the each participating practice to assist with the development of a workflow, screening process, counseling resources, and referral resources for unhealthy alcohol use. Practices in control group will receive delayed intervention at 3 months after their matched cohort of practices.
  Arms: Intervention Practices

SUMMARY:
Unhealthy alcohol use is the third leading preventable cause of death in the United States. Yet, primary care physicians do not, on average, screen for and address unhealthy alcohol use in their patient populations. By implementing practice changes to promote screening and treatment, patients stand to reduce unhealthy alcohol use and benefit from improved health outcomes. This project will provide a sample of Virginia primary care practices with a practice facilitator, practice specific resources, education on screening and counseling, and education on medication assisted therapy. The project will measure whether this change will improve screening rates and promote reduction of unhealthy alcohol use.

DETAILED DESCRIPTION:
Unhealthy alcohol use is the third leading cause of preventable death in the US. Evidence shows that screening for unhealthy alcohol use and providing persons engaged in risky drinking with brief behavioral counseling interventions improves health outcomes, collectively termed screening and brief intervention (SBI). For moderate or severe alcohol use disorder (AUD), medication assistance therapy (MAT) is effective. Despite clear evidence of effectiveness, only 13% of primary care patients are screened with a standard instrument and only 6.7% of adults with AUD receive treatment. We believe that underutilization of SBI and MAT are driven by both a misunderstanding of the role and effectiveness of primary care in addressing unhealthy alcohol and limited practice resource and infrastructure. To promote the dissemination and implementation of evidence-based strategies to address unhealthy alcohol use throughout Virginia, we have extended our EvidenceNow collaboration to include addiction medicine experts at Virginia Commonwealth University, the Virginia Ambulatory Care Outcomes Research Network (ACORN), our state's family medicine residency training programs, and our state's Community Service Boards. We propose a practice-level cluster randomized trial with wait list control. 125 primary care practices in five regions throughout the state, each centered around a residency site for educational support, will receive a practice facilitation intervention to implement screening, counseling, and treatment for unhealthy alcohol at intervention start or 6-month delay. Guided by the identified EvidenceNow key drivers for change, practice support will include practice facilitation, education and training, shared learning and best practices, screening and counseling toolkits, data support, and assessment with feedback. Each practice will identify a clinician, nurse, and administrator champion to locally lead efforts and participate in learning collaboratives. Practices will design and implement screening, counseling, and treatment processes and operational changes, adapting their implementation strategy based on experiences and findings from other sites. We will conduct a mixed methods analysis. Primary outcomes will include the increase in screening for unhealthy alcohol use, increase in provision of brief counseling interventions and MAT, and reduction in alcohol intake for patients after practices receive practice facilitation. We will use the consolidated framework for implementation research to code and rate practice facilitation (e.g. dose, mode, reach) and practice implementation strategies (e.g. SBI and MAT strategies and tools implemented) on outcomes. Data sources will include practice facilitator field notes and interviews, chart reviews, patient survey, clinician survey, All Payer Claims Data, and qualitative interviews. We will administer the patient survey at baseline, 3 months, and 6 months after the intervention. Among patients age 18 to 75 with an office visit the prior month, we will randomly select 60 to survey. In addition to our internal evaluation, we will participate in the external collaborative evaluation and dissemination activities with AHRQ throughout the project.

ELIGIBILITY:
Practice Inclusion Criteria:

1. Primary care practices
2. Ambulatory care practices

Patient Inclusion Criteria:

1. Patients 18 years and older and with an office visit at an included study site

Practice Exclusion Criteria:

1. Practices that do not provide outpatient care
2. Practices that do not provide primary care

Patient Exclusion Criteria:

1. Patients under 18 years old
2. Patients without an office visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13680 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Screening for Unhealthy Alcohol Use | 6 months
  This outcome will evaluate the percent of patients who were screened in clinic or report screening for alcohol use (numerator = intervention patients sampled who received counseling/ denominator = intervention patients who did not receive counseling at 3 time points.)
Treatment for Unhealthy Alcohol Use | 6 months
  This outcome will measure the percent of patients, screening positive for risky alcohol use, that receive any type of treatment including, but not limited to, counseling, brief intervention, motivational interviewing, referral, or medication assisted treatment.

SECONDARY OUTCOMES:
Reduction of Unhealthy Alcohol Use | 6 months
  This measure will identify the percent of patients with unhealthy alcohol use that have reduced alcohol intake after practice facilitation (numerator = number of sample patients with unhealthy alcohol use at baseline that received treatment / denominator = number of patients with unhealthy alcohol use at baseline.)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H Krist, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Virginia Ambulatory Care Outcomes Research Network, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Huffstetler AN, Villalobos G, Webel B, Rockwell MS, Funk A, Sabo RT, Epling JW, Brooks EM, Britz JB, Bortz BA, Svikis DS, Arias AJ, Tran RN, Krist AH. Practice Facilitation to Address Unhealthy Alcohol Use in Primary Care: A Cluster Randomized Clinical Trial. JAMA Health Forum. 2024 Aug 2;5(8):e242371. doi: 10.1001/jamahealthforum.2024.2371. PMID 39120895
- [Derived] Huffstetler AN, Kuzel AJ, Sabo RT, Richards A, Brooks EM, Lail Kashiri P, Villalobos G, Arias AJ, Svikis D, Bortz BA, Edwards A, Epling J, Cohen DJ, Parchman ML, Winter J, Wessler P, Yu TJ, Krist AH. Practice facilitation to promote evidence-based screening and management of unhealthy alcohol use in primary care: a practice-level randomized controlled trial. BMC Fam Pract. 2020 May 20;21(1):93. doi: 10.1186/s12875-020-01147-4. PMID 32434467

DOCUMENTS (1):
  • Informed Consent Form (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT04248023/ICF_000.pdf